CLINICAL TRIAL: NCT01883752
Title: Goal-Directed Fluid Management Based on Non- Invasive Monitoring of Pulse Oximeter-Derived Pleth Variability Index
Brief Title: Goal Directed Fluid Management Based on Non-invasive Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Maxime Cannesson, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCIANES01
Record Dates: First submitted 2012-03-07; First posted 2013-06-21 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Complication
Keywords: Goal-directed fluid therapy
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Baseline crystalloid infusion of 5 mL/kg/hr of body weight.
- Goal-directed Therapy group (Experimental): Goal-direct therapy
  Interventions: Procedure: Goal-directed Therapy group

INTERVENTIONS:
Procedure: Goal-directed Therapy group — Fluid administration is based on the respiratory variation in the pulse oximeter waveform
  Other Names: Goal Directed Fluid Optimization group
  Arms: Goal-directed Therapy group

SUMMARY:
The purpose of this study is to evaluate whether goal directed fluid management using respiratory variations in the oxygen saturation by pulse oximetry (SpO2) waveform has potential to decrease postoperative complications and outcomes.

DETAILED DESCRIPTION:
The aim of this study is to test the hypothesis that monitoring and minimizing the respiratory variations in the pulse oximeter waveform amplitude by volume loading has potential to decrease postoperative morbidity and length of stay in the hospital in patients undergoing routine, moderate-risk elective surgery.

In this study the investigators will test the impact of hemodynamic optimization based on the respiratory variations in the plethysmographic waveform amplitude to decrease postoperative morbidity and length of stay in the hospital in patients undergoing routine, moderate-risk elective surgery. The primary outcome variable is the incidence of postoperative complications. Secondary outcome variables are the duration of hospital and ICU stays, postoperative mortality, and cost of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female)
* Over 18 years old undergoing non-cardiac surgery
* Weight > 40 kg, Body Mass Index < 40

Exclusion Criteria:

* Patients who do not consent
* Body Mass Index > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | Maximum 90 days after surgery
  The length of stay in the hospital is defined as postoperative number of days in the hospital until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Cannesson, MD, PhD, Principal Investigator — UC Irvine Medical Center, Dept of Anesthesiology & Perioperative Care
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Bennett-Guerrero E, Welsby I, Dunn TJ, Young LR, Wahl TA, Diers TL, Phillips-Bute BG, Newman MF, Mythen MG. The use of a postoperative morbidity survey to evaluate patients with prolonged hospitalization after routine, moderate-risk, elective surgery. Anesth Analg. 1999 Aug;89(2):514-9. doi: 10.1097/00000539-199908000-00050. PMID 10439777
- [Background] Mythen MG, Webb AR. Intra-operative gut mucosal hypoperfusion is associated with increased post-operative complications and cost. Intensive Care Med. 1994;20(2):99-104. doi: 10.1007/BF01707662. PMID 8201106
- [Background] Chappell D, Jacob M, Hofmann-Kiefer K, Conzen P, Rehm M. A rational approach to perioperative fluid management. Anesthesiology. 2008 Oct;109(4):723-40. doi: 10.1097/ALN.0b013e3181863117. PMID 18813052
- [Background] Lebuffe G, Vallet B, Takala J, Hartstein G, Lamy M, Mythen M, Bakker J, Bennett D, Boyd O, Webb A. A european, multicenter, observational study to assess the value of gastric-to-end tidal PCO2 difference in predicting postoperative complications. Anesth Analg. 2004 Jul;99(1):166-72. doi: 10.1097/00000539-200407000-00034. PMID 15281524
- [Background] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Background] Venn R, Steele A, Richardson P, Poloniecki J, Grounds M, Newman P. Randomized controlled trial to investigate influence of the fluid challenge on duration of hospital stay and perioperative morbidity in patients with hip fractures. Br J Anaesth. 2002 Jan;88(1):65-71. doi: 10.1093/bja/88.1.65. PMID 11881887
- [Background] Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, Fleming SC. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. Br J Anaesth. 2005 Nov;95(5):634-42. doi: 10.1093/bja/aei223. Epub 2005 Sep 9. PMID 16155038
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Conway DH, Mayall R, Abdul-Latif MS, Gilligan S, Tackaberry C. Randomised controlled trial investigating the influence of intravenous fluid titration using oesophageal Doppler monitoring during bowel surgery. Anaesthesia. 2002 Sep;57(9):845-9. doi: 10.1046/j.1365-2044.2002.02708.x. PMID 12190747
- [Background] Poeze M, Greve JW, Ramsay G. Meta-analysis of hemodynamic optimization: relationship to methodological quality. Crit Care. 2005;9(6):R771-9. doi: 10.1186/cc3902. Epub 2005 Nov 15. PMID 16356226